CLINICAL TRIAL: NCT01386307
Title: ¿Cuál es la Prevalencia de Dolor en internación en el Hospital Italiano?
Brief Title: Prevalence of Pain in Inpatient at the Hospital Italiano de Buenos Aires
Acronym: Pain
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1670
Record Dates: First submitted 2011-05-27; First posted 2011-07-01 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pain
Keywords: Pain; Hospitalization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the prevalence of patients with acute and chronic pain in the area of inpatient at the Hospital Italiano de Buenos Aires.

DETAILED DESCRIPTION:
The diagnosis and treatment of pain during hospitalization are becoming increasingly important. In recent decades there have been articles that explain that pain is underdiagnosed, that there are patients who do not receive treatment or that it fails to decrease pain intensity. It has now been shown that pain is a common problem during hospitalization, showing a prevalence of 38 to 91% depending on the population studied.

Published studies show that there are three types of pain during hospitalization: acute or chronic pain that motivates the admission and continues during hospitalization, pain that appears during hospitalization but was not the cause of the admission or associated with health care, and,pain that appears during the hospitalization associated with health care. To complete the description of patients with pain during hospitalization it has been suggested the existence of a fourth group of patients presenting with chronic pain that does not motivate the admission but persists and does not interfere during hospitalization. In a study evaluating the Italian population shows that the prevalence of pain is modified by marital status and age, and the intensity of pain increases with time evolution of pain and days of hospital stay. Some studies, mainly in Europe, show that the use of analgesics is high but the adherence to guideline recommendations for treatment of pain is low, or that the presence of pain is not recorded in the medical chart compared to the indication of analgesic treatment.

These results demonstrate the need to determine the prevalence of pain in hospitalization at each institution, distinguishing the case of pain prior to admission or appearing during the same (or motivation), evaluating the indication of pain at each hospital, in order to learn about the current situation and design and implement actions to improve pain management in this institution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years.
* Evaluated at 48 hours after hospital admission in areas general hospitalization, coronary care unit, adult intensive care, intermediate care and day hospital of the Hospital Italiano Central

Exclusion Criteria:

* Refusal to participate in the study or the informed consent process.
* Inability to understand or express pain (aphasia, dementia).
* Alteration ef the sensory.
* Language other than Spanish.
* Inpatient at the emergency room.
* Presence of acute confusion or delirium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years, hospitalized at the Hospital Italiano de Buenos Aires and admitted 24 to 72 hours before the evaluation.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of pain | within 48 to 72 hours after admission to hospital
  Presence of pain in the last 24 hours of hospitalization

SECONDARY OUTCOMES:
Response to analgesic treatment | within 48 to 72 hours after admission to hospital
The cause of pain during hospitalization | within 48 to 72 hours after admission to hospital
Number of patients reporting pain to heath care personnel | within 48 to 72 hours after admission to hospital
Proportion of physicians who know the patient is in pain according to the evolution in medical chart | within 48 to 72 hours after admission to hospital
Number of nurses who know that the patient has pain according to medical chart | within 48 to 72 hours after admission to hospital
Proportion of hospitalized patients treated for pain | within 48 to 72 hours after admission to hospital
Type of analgesic treatment received | within 48 to 72 hours after admission to hospital
Number of patients with pain evaluated by a pain specialist | within 48 to 72 hours after admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Diego Giunta, MD, Study Director — Hospital Italiano de Buenos Aires; Maria L Bechelli, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Jimena Vicens, MD, Study Chair — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad de Buenos Aires, Buenos Aires, Argentina